CLINICAL TRIAL: NCT03266341
Title: Detection of Anaerobes in Different Clinical Samples
Brief Title: Detection of Anaerobes in Different Clinicalsamples
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Safaa Samir, Detection of anaerobes in different clinical samples, Assiut University
Other Study IDs: Anaerobes detection in samples
Record Dates: First submitted 2017-08-28; First posted 2017-08-30 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Anaerobic Bacterial Infection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Cultures — Take different samples anddetection of anaerobes on enriched blood agar and other selective anaerobic cultures

SUMMARY:
Early detection of anaerobic bacteria to avoid its serious comlications

DETAILED DESCRIPTION:
Infections caused by anaerobic bacteria are common and may be serious and life-threatening.Obligately anaerobic bacteria do not grow on solid media in room air (0.04% carbon dioxide and 21% oxygen); facultatively anaerobic bacteria can grow in the presence or absence of air. Microaerophilic bacteria do not grow at all aerobically or grow poorly, but grow better under 10% carbon dioxide or anaerobically. Anaerobic bacteria can be divided into strict anaerobes that can not grow in the presence of more than 0.5% oxygen and moderate anaerobic bacteria that are able of growing between 2 and 8% oxygen. Anaerobic bacteria usually do not possess catalase, but some can generate superoxide dismutase which protects them from oxygen.

Anaerobes are the predominant components of the bacterial flora of normal human skin and mucous membranes, and are therefore a common cause of bacterial infections of endogenous origin. Infections due to anaerobic bacteria can evolve all body systems and sites . The predominant ones include: abdominal, pelvic, respiratory, and skin and soft tissues infections. Because of their fastidious nature, they are difficult to isolate from infectious sites and are often overlooked. Failure to direct therapy against these organisms often leads to clinical failures. Their isolation requires appropriate methods of collection, transportation, and cultivation of specimens. Treatment of anaerobic bacterial infection is complicated by the slow growth of these organisms, which makes diagnosis in the laboratory possible only after several days, by their often polymicrobial nature and by the growing resistance of anaerobic bacteria to antimicrobial agent.

Almost all anaerobic infections originate from the patient's own microflora. Poor blood supply and tissue necrosis lower the oxidation-reduction potential and favor the growth of anaerobes. Any condition that lowers the blood supply to an affected area can predispose to anaerobic infection. Therefore, foreign body, malignancy, surgery, edema, shock, traum and vascular disease may predispose to anaerobic infection. Previous infection with aerobic or facultative organisms also may make the local tissue conditions more favorable for the growth of anaerobic organisms. The human defense mechanisms also may be impaired by anaerobic conditions .

ELIGIBILITY:
Inclusion Criteria:

- Patient with infection organism not yet detected

Exclusion Criteria:

* patients with infection organism is already detected

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Take different samples for dtection of the causitive anaerobe
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-09-15 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Detection of anaerobes in different clinical samples | 2years
  Samples will be in oculated on different anaerobic media

CONTACTS AND LOCATIONS:
Overall Officials: Sohair Mohamed ahmed, Proffisor, Study Director — Proffisor; Asmaa Omar ahmef, Assistant prof, Principal Investigator — Assistant pro